CLINICAL TRIAL: NCT06247215
Title: Development of a Culturally Tailored Resilience-Building Intervention to Facilitate Advance Care Planning Discussions Between Chinese American Patients and Their Family Caregivers
Brief Title: Building Resilience for Advance Care Planning (ACP) in Chinese Americans
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Chicago (Other); Rush University Medical Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2023-0354; P50MD017349 (NIH)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Religious Leaders: Religious leaders providing spiritual care to Chinese Americans
  Interventions: Other: Religious leaders
- Chinese Americans living in Chicago: Chinese Americans living in Chicago
  Interventions: Other: Chinese Americans
- Chinese Americans for end-of-life care discussions: Chinese Americans with experience in end-of-life care discussions
  Interventions: Other: Chinese Americans with end-of-life care discussions
- Chinese Americans with chronic disease and their family members: Chinese Americans diagnosed with cancer, hypertension, or heart disease and their family members
  Interventions: Other: Chinese Americans with chronic diseases

INTERVENTIONS:
Other: Religious leaders — Religious leaders who have experience providing pastoral or spiritual care to Chinese Americans living in Chicago
  Groups: Religious Leaders
Other: Chinese Americans — Chinese Americans living in Chicago.
  Groups: Chinese Americans living in Chicago
Other: Chinese Americans with end-of-life care discussions — Chinese Americans who have experience discussing end-of-life care decisions with others.
  Groups: Chinese Americans for end-of-life care discussions
Other: Chinese Americans with chronic diseases — Chinese Americans who are diagnosed with cancer, hypertension, or heart disease and their family caregivers
  Groups: Chinese Americans with chronic disease and their family members

SUMMARY:
The goal of this observational study is to learn about how Chinese Americans engage in advance care planning (ACP) discussions with their family caregivers.

The main questions it aims to answer are:

1. How do religious leaders discuss advance care planning and death-related topics with Chinese Americans who are diagnosed with cancer or heart disease in Chicago?
2. Are Chinese Americans living in Chicago ready to participate in ACP discussions with their family?
3. What kind of support and resources are required to engage in end-of-life care discussions among Chinese Americans/immigrants living in Chicago?
4. What do Chinese Americans with cancer, high blood pressure, or heart disease and their family members think about an ACP pamphlet made for Chinese Americans?

Participants will share their experience either through interviews or a survey.

DETAILED DESCRIPTION:
The overall objective of this pilot study is to develop a culturally tailored resilience-building intervention for Chinese Americans with cancer or heart disease in Chicago. A qualitative analysis of semi-structured interviews will be conducted to identify how religious leaders addressed death-related topics with Chinese Americans with cancer, heart disease, or hypertension in Chicago. In addition, a mixed-method study using surveys and focus groups to understand the readiness, support, and resources of Chinese Americans living in Chicago to participate in ACP discussions with their family. Finally, a usability study will ask Chinese Americans with cancer, high blood pressure, or heart disease, and their family members, to share feedback on an ACP pamphlet designed for Chinese Americans.

ELIGIBILITY:
Group 1

Inclusion criteria for religious leaders:

* Age ≥ 18 years of age;
* Having served as a chaplain, pastor, or monk at a health care setting or religious organization in Chicago;
* Being able to read and respond to questions in English or Mandarin;
* Having experience in having end-of-life discussions with Chinese Americans in Chicago.

Exclusion criteria: Unwilling to provide consent.

Group 2

Inclusion criteria for Chinese Americans living in Chicago:

* Age ≥ 18 years of age;
* Identifying themselves as first- or second-generation Chinese Americans;
* Being able to read and respond to questions in Mandarin or English.

Exclusion criteria: Unwilling to provide consent.

Group 3

Inclusion criteria for Chinese Americans with experience in end-of-life care discussions:

* Age ≥ 18 years of age;
* Identifying themselves as first- or second-generation Chinese Americans;
* Having experience discussing end-of-life care decisions with others;
* Being able to read, write, and respond to questions in either English or Mandarin.

Exclusion criteria: Unwilling to provide consent.

Group 4

Inclusion criteria for Chinese Americans with cancer, hypertension, or heart disease:

* Age ≥ 18 years of age;
* Self-identify themselves as first- or second-generation Chinese Americans/immigrants;
* Having a diagnosis of chronic diseases, such as cancer, hypertension, or heart disease;
* Being able to read and respond to questions in Mandarin;
* Being of the non-Hispanic Asian race/ethnicity.

Exclusion criteria:

* Having cognitive impairment per a Short Portable Mental Status Questionnaire with more than 3 errors, or
* Being born in the US.

Inclusion criteria for their family members:

* Age ≥ 18 years of age;
* Being able to read and respond to questions in Mandarin;
* Having a family member who is self-identified as a first or second-generation Chinese American/immigrant and has been diagnosed with chronic diseases, such as cancer, hypertension, or heart disease.

Exclusion criteria: Unwilling to provide consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have experience providing spiritual/pastoral care to Chinese Americans in Chicago as a chaplain, pastor, or monk at a health care setting or religious organization in Chicago, or who self-identify as first- or second-generation Chinese Americans living in Chicago with/without having end-of-life care discussions with others. Chinese Americans living with cancer, hypertension, or heart disease, and their family members
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Readiness, Support and Resources for ACP Discussions | Immediately at the end of the study
  The Advance Care Planning Engagement Survey was used to evaluate the readiness for advance care planning discussions among Chinese Americans living in Chicago.

SECONDARY OUTCOMES:
Support Needed for ACP Discussions | Immediately at the end of the study
  An in-depth understanding of the support and resources needed to engage in ACP discussions with their family among Chinese Americans who have experience discussing end-of-life care with others.
Strategies Used for ACP and Death-related Discussions | Immediately at the end of the study
  An in-depth understanding of barriers and strategies used to assist Chinese Americans/immigrants in ACP and death-related discussions.
Acceptability of an ACP pamphlet | Immediately at the end of the study
  An in-depth understanding of Chinese Americans' views and acceptability on an ACP pamphlet.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States